CLINICAL TRIAL: NCT04481854
Title: Cricoid Pressure Versus Paratracheal Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of the anesthesia and intensive care department, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Sellick vs paratracheal
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cricoid Pressure During Tracheal Intubation
Keywords: cricoid pressure; paratracheal pressure

STUDY DESIGN:
Intervention Model Description: patients will be randomized to recieve cricoid pressure or left paratracheal pressure
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cricoid pressure group (Experimental): Patients of this group will recieve cricoid pressure during direct laryngoscopy.
  Interventions: Procedure: cricoid pressure
- left paratracheal pressure group (Experimental): Patients of this group will recieve left paratracheal pressure during direct laryngoscopy.
  Interventions: Procedure: left paratracheal pressure

INTERVENTIONS:
Procedure: cricoid pressure — cricoid pressure during laryngoscopy
  Arms: Cricoid pressure group
Procedure: left paratracheal pressure — left paratracheal pressure during laryngoscopy
  Arms: left paratracheal pressure group

SUMMARY:
Prospective randomized trial, including adult patients scheduled for orthopedic or abdominal surgery under general anesthesia and tracheal intubation. in this study the investigators will compare the classic cricoid pressure and the left paratracheal pressure regarding their impact on the intubation condition and the effectiveness.

DETAILED DESCRIPTION:
Prospective randomized trial, including adult patients scheduled for orthopedic or abdominal surgery under general anesthesia and tracheal intubation. in this study the investigators will compare the classic cricoid pressure and the left paratracheal pressure regarding their impact on the intubation condition and the effectiveness.

During the laryngoscopy, the modification of the Cormack and Lehane grade before and after the application of the cricoid or paratracheal pressure will be noticed.

concerning the effectiveness of the procedure, a gastric tube will be introduced through the oesophagus during the procedure, under direct vision.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with no criteria of difficult intubation or mask ventilation
* no criteria of full stomach requiring crush induction

Exclusion Criteria:

* Unexpected difficult laryngoscopy or mask ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Modification of Cormack and Lehane grade | 3 minutes after induction of general anesthesia
  Cormack and Lehane grade before and after the procedure

SECONDARY OUTCOMES:
Effectiveness of the pressure | 5 minutes after induction of general anesthesia
  Possibility to introduce a gastric tube through the oesophagus

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No